CLINICAL TRIAL: NCT01042860
Title: The Influence of Lutein Supplements on Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Cognis Deutschland GmbH & Co. KG (Industry)
Responsible Party: Dr. Christine Gärtner, Cognis Deutschland GmbH & Co. KG
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 061052
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Age-Related Macular Degeneration
Keywords: macular pigment; lutein; age-related macular degeneration; AMD
MeSH Terms: conditions — Macular Degeneration | interventions — Lutein

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- supplement (Active Comparator): lutein supplement
  Interventions: Dietary Supplement: Lutein
- placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lutein — Lutein supplement, 10 mg daily
  Arms: supplement
Dietary Supplement: Placebo — Placebo
  Arms: placebo

SUMMARY:
Rationale: Age-related macular degeneration is the most common cause of blindness in the industrialized world. Macular pigment is hypothesized to protect against the vision loss in this disease.

Objective: 1. To study if the macular pigment optical density can be raised by lutein supplementation. 2. To study if lutein supplementation can stop or slow down the decrease in visual functions.

Study design: Randomized, double blind, placebo controlled intervention study.

Study population: Eighty patients with early signs of age-related macular degeneration Intervention: The intervention group (40 subjects) receives 10 mg lutein per day, while the control group (40 subjects) gets a placebo.

ELIGIBILITY:
Inclusion Criteria:

* AMD grade 2 or 3
* visual acuity > 0.5
* BMI < 30

Exclusion Criteria:

* using lutein supplements
* smoking
* diabetes
* diseases that interfere with lipid absorption
* other eye diseases

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Macular Pigment Optical Density | Baseline, 4 months, 8 months, 12 months

SECONDARY OUTCOMES:
Visual Acuity | Baseline, 4 months, 8 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tos TJM Berendschot, PhD, Principal Investigator — University Eye Clinic Maastricht; Ian J Murray, PhD, Principal Investigator — University of Manchester
Locations (2):
- University Eye Clinic Maastricht, Maastricht, Netherlands
- Faculty of Life Sciences, University of Manchester, Manchester, United Kingdom

REFERENCES:
- [Derived] Murray IJ, Makridaki M, van der Veen RL, Carden D, Parry NR, Berendschot TT. Lutein supplementation over a one-year period in early AMD might have a mild beneficial effect on visual acuity: the CLEAR study. Invest Ophthalmol Vis Sci. 2013 Mar 11;54(3):1781-8. doi: 10.1167/iovs.12-10715. PMID 23385792